CLINICAL TRIAL: NCT06091449
Title: The Effect of High Fidelity and Virtual Reality-Based Simulation Applications on Simulation-Based Learning, Reflective Thinking and Therapeutic Communication Skills in Undergraduate Nursing Students
Brief Title: High Fidelity Simulation and Virtual Reality and Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe ARIKAN DÖNMEZ, associate professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-66777842-000-00003054201
Record Dates: First submitted 2023-09-18; First posted 2023-10-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Nursing Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fidelity simulation (Experimental): The Faculty of Nursing has a simulation laboratory to enable students to realize their professional skills in a high-reality environment. The laboratory has all the equipment that should be found in a clinic, such as a high-reality simulation mannequin, nurse's table, patient bed, shelves, monitors, bedside oxygen systems, treatment and emergency response carts.Lab; It consists of 3 sections: application room, control room and analysis room.
  Interventions: Other: High fidelity simulation
- High fidelity simulation and virtual reality (Experimental): The modular education and virtual reality-based simulation program is currently actively available on the "hadi.hacettepe.edu.tr" website. Students who will benefit from this program can access the program after defining a username and password.The application of high-fidelity simulation is the same in both groups.
  Interventions: Other: High fidelity simulation; Other: Virtual reality

INTERVENTIONS:
Other: High fidelity simulation — Within the scope of high reality simulation application; The ideal number of students to take part in each simulation was determined to be 10. On the simulation day, the researchers responsible for the simulation application will introduce the environment and the tools and equipment they will use in the simulation application, so that they can make preliminary preparations for the students. It will last 60 minutes in total, including preliminary information (10 minutes), simulation time (15 minutes) and evaluation/analysis session (35 minutes).
Other: Virtual reality — For the virtual reality-based simulation application, students can log in to the virtual reality-based simulation program prepared in line with the "Diabetes Mellitus" scenario using their username and password; They will receive modular training integrated into the simulation. The expected time for students to complete the modular training is 30 minutes. Students who complete the module will be asked to take a 10-minute break and then participate in a virtual reality-based simulation application.The application of high-fidelity simulation is the same in both groups.
  Arms: High fidelity simulation and virtual reality

SUMMARY:
Subject:

The effects of high fidelity and virtual reality-based simulation applications on simulation-based learning, reflective thinking and therapeutic communication skills in nursing undergraduate students.

Objective : It was planned to determine the effects of high fidelity and virtual reality-based simulation applications on simulation-based learning, reflective thinking and therapeutic communication skills in nursing undergraduate students.

Backgroud:Simulation-based learning is one of the most effective and interesting teaching methods that is effective in adapting nursing students to clinical environments by reducing the gap between education and practice.Students reinforce their knowledge and improve their clinical performance through active training methods that mimic real healthcare environments. They have the experience of developing psychomotor skills and making appropriate decisions in a timely manner through supervision, repetition and reinforcement.

Methods:The research is planned to be conducted at Hacettepe University Faculty of Nursing between 16 October 2023 and 16 October 2024.Students will be divided into two groups by randomization method. The group that will receive virtual reality application is 38 people; The group for which simulation + virtual reality application will be applied will be determined as 38 people.Data will be collected using the Personal Information Form, simulation-based learning evaluation scale, reflective thinking skills scale for problem solving, and therapeutic communication skills scale for nursing students.The analysis of the data will be done with a statistical program.

DETAILED DESCRIPTION:
Place of the research The research was planned to be carried out at Hacettepe University Faculty of Nursing. Scenarios will be based on diabetes mellitus so that the case topics to be managed in high fidelity and virtual reality-based simulation applications are equivalent. Nursing the faculty has a simulation laboratory to enable students to realize their professional skills in a high- fidelity environment. The laboratory has all the equipment that should be found in a clinic, such as a high- fidelity simulation mannequin, nurse's table, patient bed, shelves, monitors, bedside oxygen systems, treatment and emergency response carts. Lab; It consists of 3 sections: application room, control room and analysis room. As a result of the Research Infrastructure Project (No: TAY-2022-19754) supported by Hacettepe University Scientific Research Projects Coordination Unit, virtual reality-based simulation will be available as of 2023. Program is located in the infrastructure of the faculty of nursing. This program includes 3 different modular training on the topics of "Diabetes Mellitus", "Chemotherapy Treatment" and "Dementia" and virtual reality-based simulation scenarios for these topics. The modular education and virtual reality-based simulation program is currently actively available on the "hadi.hacettepe.edu.tr" website. Students who will benefit from this program can access the program after defining a username and password. The content of the module on the subject of "Diabetes Mellitus" within the scope of this program; It includes topics such as the definition of dementia, risk factors, signs and symptoms, complications, treatment and nursing care, and patient and/or caregiver education. Learning activities such as question and answer applications and gamification are also included to keep students active during the education process and to make interim evaluations. There are. After applying the Diabetes Mellitus module, students complete the program by switching to a virtual reality-based simulation program for Diabetes Mellitus. They will also implement a virtual reality-based interactive therapeutic diabetes mellitus patient education program here.

Universe of Research The universe of the research; It will consist of second-year students studying at Hacettepe University Faculty of Nursing in the 2023-2024 academic year. The main purpose of selecting this student group is that it is a group of students who have successfully completed the Nursing Fundamentals course in the second year, have basic knowledge and skills in nursing care, but are still not sufficiently equipped to intervene with the patient. While this student group is still at the beginning of education and applications, it is thought that by determining the effect of simulation applications based on high fidelity and virtual reality, it will raise awareness in this field and the use of this method in the following educational processes will make significant contributions to student education.

Sample of the Research G*Power-3.1.9.4 program was used to calculate the sample size and power of the study. Accordingly, taking α = 0.05 (Type I error), each test was determined at 85% power and 5% significance level. It was planned to complete the research with a total of 68 students, 34 in a group. Considering possible 10% data loss, the research was planned to be completed with 76 students. The group that will receive virtual reality application is 38 people; The group for which simulation + virtual reality application will be applied will be determined as 38 people.

Preparation of Data Collection Form In the research, data will be collected with the following tools. PRE-TESTS include personal information form, simulation-based learning evaluation scale, reflective thinking skill scale for problem solving, therapeutic communication skills scale for nursing students; POST TESTS include the simulation-based learning assessment scale, the reflective thinking skill scale for problem solving, and the therapeutic communication skills scale for nursing students.

Collection of Data Students who meet the inclusion criteria and agree to participate in the research will be informed, and any questions they have about the operation of the research will be answered. It will be explained during the interview that the information collected will not be stated or published in the research and will be kept as a record. The Voluntary Participation form will be explained, they will be asked to read the consent form, give their consent voluntarily and it will be recorded. Data will be collected through forms and scales hand-delivered to students by the researchers.

Application of Research An introduction and information meeting will be held before the research for students who meet the research criteria and agree to participate in the study. Written informed consent of the students will be obtained. Face-to-face information about the research was given to the participants who will be included in the research.After being informed, they will be asked to fill out the Personal Information Form, the simulation-based learning evaluation scale, the reflective thinking skill scale for problem solving, and the therapeutic communication skills scale for nursing students in order to complete the PRE-TESTS. Following the completion of the Pretests, participants will be assigned to one of two groups, Group-1 (high fidelity simulation application) and Group-2 (high fidelity and virtual reality based simulation application), according to the block randomization method to be carried out in a computerized environment.

Evaluation of Data The data obtained from the research will be evaluated by transferring it to IBM SPSS (Statistical Packages for the Social Sciences) Statistics 23 program. When evaluating the data, descriptive statistics (mean, standard deviation, median, minimum, maximum) will be used for continuous variables and frequency distribution will be used for categorical variables. Differences between categorical variables were evaluated using Chi-square test and Fisher Exact test, numerical variables were evaluated using Chi-square test and Fisher Exact test.

The relationships between them will be evaluated with Spearman Correlation Analysis. The suitability of the data for normal distribution will be evaluated with the Shapiro Wilk normality test and Q-Q graphs. Accordingly, if the parametric test assumptions are met, the Significance Test of the Difference Between Two Means is used to compare independent group differences; When parametric test assumptions cannot be met, the Mann-Whitney U test will be used.

In dependent group comparisons, if parametric test assumptions are met, Repeated Measurements Variance Analysis and Significance Test of the Difference Between Two Spouses; When parametric test assumptions are not met, Friedman Test and Wilcoxon Paired Two Sample Test will be used.

In all analyses, a p value of ≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being a second year student at the Faculty of Nursing
* Being 18 years or older
* Voluntarily agreeing to participate in the research
* have internet access
* Not having participated in high reality and/or virtual reality based applications before

Exclusion Criteria:

* Not participating in any of the pretest-posttest tests
* Not agreeing to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Simulation Based Learning Scale | Change from baseline scores at the end of 60 minutes.
  It evaluates the simulation-based learning experience from the student perspective. The scale has 5 sub-dimensions and 37 items. The responses are scored on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) and the total score ranges between 37-185. All statements in the scale are positive and there are no reverse coded items. It will be applied to the students just before high reality simulation and/or virtual reality simulation and after completing the training on the same day (each session is 60 minutes).
Reflective Thinking Skills for Problem Solving Scale | Change from baseline scores at the end of 60 minutes.
  It evaluates reflective thinking towards problem solving. It is a 5-point Likert scale (Always=5, Most of the time=4, Sometimes=3, Rarely=2, Never time=1) and consists of 14 items. The highest score to be obtained from the scale is 70 and the lowest score is 14. The maximum score is expressed as the degree of having reflective thinking skills. It will be applied to the students just before high reality simulation and/or virtual reality simulation and after completing the training on the same day (each session is 60 minutes).
Therapeutic Communication Skills Scale | Change from baseline scores at the end of 60 minutes.
  It measures nursing students' therapeutic communication skills. It consists of 3 dimensions, 16 It is a 7-point Likert-type scale consisting of items. Scores to be obtained from the scale range from 16-112. An increase in the score indicates an increase in therapeutic communication skills. It will be applied to the students just before high reality simulation and/or virtual reality simulation and after completing the training on the same day (each session is 60 minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No